CLINICAL TRIAL: NCT07165951
Title: A Randomized, Double-blind, Parallel-controlled, Multicenter Phase III Clinical Trial Comparing TQB2868 Injection Combined With Anlotinib Hydrochloride Capsules to Placebo Combined With Chemotherapy as First-line Treatment for Metastatic Pancreatic Ductal Adenocarcinoma (mPDAC)
Brief Title: Clinical Trial Comparing TQB2868 Injection Combined With Anlotinib Hydrochloride Capsules With Placebo Combined With Chemotherapy as First-line Treatment for Metastatic Pancreatic Ductal Adenocarcinoma (mPDAC)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Chia Tai Tianqing Pharmaceutical Technology Development Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TQB2868-ALTN-III-01
Record Dates: First submitted 2025-09-03; First posted 2025-09-10 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-06

CONDITIONS: Metastatic Pancreatic Ductal Adenocarcinoma
MeSH Terms: interventions — Gemcitabine; Paclitaxel; Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TQB2868 Injection+Anlotinib Hydrochloride Capsules+chemotherapy (Experimental): TQB2868 Injection+Anlotinib Hydrochloride Capsules+Gemcitabine Hydrochloride Injection+Paclitaxel for Injection
  Interventions: Drug: TQB2868 Injection; Drug: Anlotinib Hydrochloride Capsules; Drug: Gemcitabine Hydrochloride Injection; Drug: Paclitaxel for Injection
- TQB2868 Placebo+Anlotinib Hydrochloride Capsules+chemotherapy (Placebo Comparator): TQB2868 Placebo+Anlotinib Hydrochloride Capsules+Gemcitabine Hydrochloride Injection+Paclitaxel for Injection
  Interventions: Drug: Anlotinib Hydrochloride Capsules; Drug: Gemcitabine Hydrochloride Injection; Drug: Paclitaxel for Injection; Drug: TQB2868 Placebo

INTERVENTIONS:
Drug: TQB2868 Injection — TQB2868 injection: PD-L1 and Transforming Growth Factor-beta (TGF - β) dual antibody
  Arms: TQB2868 Injection+Anlotinib Hydrochloride Capsules+chemotherapy
Drug: Anlotinib Hydrochloride Capsules — Anlotinib Hydrochloride Capsules
Drug: Gemcitabine Hydrochloride Injection — Gemcitabine Hydrochloride Injection
Drug: Paclitaxel for Injection — Paclitaxel for Injection
Drug: TQB2868 Placebo — TQB2868 Placebo without drug substance
  Arms: TQB2868 Placebo+Anlotinib Hydrochloride Capsules+chemotherapy

SUMMARY:
This study adopts a randomized, open label, placebo-controlled, multicenter trial design. OS was the primary endpoint, and eligible subjects were randomly divided into 1:1 groups and received TQB2868 injection and anlotinib hydrochloride capsules combined with chemotherapy, compared to placebo combined with chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. The subjects voluntarily joined this study, signed the Informed Consent Form (ICF), and showed good compliance;
2. On the date of signing the ICF, aged between 18 and 75 years old (inclusive);
3. Pancreatic ductal adenocarcinoma (PDAC) diagnosed by tissue or cytology;
4. According to the American Joint Commission on Cancer (AJCC) 8th Edition Tumor, Node, Metastasis (TNM) staging system for pancreatic cancer, patients with stage IV metastatic pancreatic cancer;
5. Have not received any systemic anti-tumor treatment or investigational drug therapy; If receiving neoadjuvant/adjuvant therapy, the time interval between the last administration and recurrence/progression must be ≥ 6 months, and the toxicity related to anti-tumor therapy has recovered to ≤ level 1 or the toxicity level specified in the inclusion criteria (excluding hair loss); According to RECIST v1.1, there is at least one measurable lesion. If the lesion has undergone local treatment (radiotherapy, ablation, interventional therapy, etc.) in the past, it must be clearly proven to have progressed in accordance with RECIST v1.1 before it can be considered a measurable lesion;

7. Eastern Cooperative Oncology Group (ECOG) score from 0 to 1; Expected survival is greater than 12 weeks; 9. The laboratory inspection meets the protocol standards; 10. Women of childbearing age should agree to use effective contraceptive measures during the study period and within 6 months after the end of the study, and have a negative serum test within 7 days before enrollment in the study; Men should agree to use effective contraceptive measures during the study period and within 6 months after the end of the study period;

Exclusion Criteria:

1. Have had or currently have other malignant tumors within the past 5 years prior to the first use of medication;
2. There are various factors that affect intravenous injection, venous blood collection diseases, or oral medication (such as inability to swallow, chronic diarrhea, and intestinal obstruction);
3. Adverse reactions from previous treatments have not recovered to NCI CTCAE v5.0 score ≤ 1, except for toxicity that has been determined by researchers to have no safety risks, such as grade 2 hair loss, grade 2 peripheral neurotoxicity, non clinically significant, and asymptomatic laboratory abnormalities;
4. Those who have received major surgical treatment, significant traumatic injury, or are expected to undergo major surgery during the expected study treatment period within 4 weeks before the first medication, or have long-term untreated wounds or fractures;
5. Subjects who experience any bleeding or bleeding events ≥ NCI CTCAE v5.0 grade 3 within 4 weeks prior to the first administration;
6. Individuals who have experienced arterial/venous thrombotic events within 6 months prior to the first administration, such as cerebrovascular accidents (including transient ischemic attacks), deep vein thrombosis, pulmonary embolism, or any other history of severe thromboembolism (implantable venous infusion port or catheter-related thrombosis, or superficial vein thrombosis is not considered "severe" thromboembolism);
7. hepatitis B virus (HBV) infected individuals cannot receive regular antiviral treatment throughout the entire process; HCV infected individuals (HCV Ab or HCV RNA positive): Researchers determine that they are in an unstable state or need to continue antiviral treatment. Regular antiviral treatment cannot be accepted during the study;
8. Active syphilis infected individuals who require treatment;
9. History of active pulmonary tuberculosis, idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonia, radiation pneumonitis requiring treatment, or clinically symptomatic active pneumonia;
10. Individuals with a history of abuse of psychotropic drugs who are unable to quit or have mental disorders;
11. Individuals who are preparing for or have previously undergone allogeneic bone marrow transplantation or solid organ transplantation;
12. Subjects with any severe and/or uncontrolled illnesses;
13. Subjects who require immunosuppressive therapy, systemic or absorbable local hormone therapy to achieve immunosuppression and continue to use it within 7 days prior to the first dose (excluding corticosteroids with a daily dose of<10 mg prednisone or other therapeutic hormones);
14. Tumor related symptoms are difficult to control;
15. Known to be allergic to the components of research drug excipients;
16. Those who have participated in and used other anti-tumor clinical trial drugs within 4 weeks before the first medication;
17. Pregnant or breastfeeding subjects; According to the judgment of the researchers, there are serious situations that pose a threat to the safety of the subjects or affect their ability to complete the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 566 (Estimated)
Dates: Start 2025-12-02 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | The duration is approximately 2 years
  By evaluating overall survival (OS), this study aims to demonstrate the efficacy of TQB2868 injection combined with anlotinib hydrochloride capsules in chemotherapy compared to placebo combined with chemotherapy in the first-line treatment of metastatic pancreatic ductal adenocarcinoma (mPDAC).

SECONDARY OUTCOMES:
Progression-Free Survival evaluated by researchers | The duration is approximately 1 year
  Evaluate the effectiveness of TQB2868 injection and anlotinib hydrochloride capsules combined with chemotherapy compared to placebo combined with chemotherapy in first-line treatment of metastatic pancreatic ductal adenocarcinoma (mPDAC) using the Progression-Free Survival evaluated by researchers.
Objective Response Rate evaluated by researchers | The duration is approximately 1 year
  Evaluate the effectiveness of TQB2868 injection and anlotinib hydrochloride capsules combined with chemotherapy compared to placebo combined with chemotherapy in first-line treatment of metastatic pancreatic ductal adenocarcinoma (mPDAC) using the Objective Response Rate evaluated by researchers.
The Disease Control Rate evaluated by the researchers | The duration is approximately 1 year
  Evaluate the effectiveness of TQB2868 injection and anlotinib hydrochloride capsules combined with chemotherapy compared to placebo combined with chemotherapy in first-line treatment of metastatic pancreatic ductal adenocarcinoma (mPDAC) using the Disease Control Rate evaluated by researchers.
The Duration of Response (DOR) evaluated by the researchers | The duration is approximately 1 year
  Evaluate the effectiveness of TQB2868 injection and anlotinib hydrochloride capsules combined with chemotherapy compared to placebo combined with chemotherapy in first-line treatment of metastatic pancreatic ductal adenocarcinoma (mPDAC) using the Duration of Response evaluated by researchers.
The Time to Tumor Recurrence evaluated by the researchers | The duration is approximately 1 year
  Evaluate the effectiveness of TQB2868 injection and anlotinib hydrochloride capsules combined with chemotherapy compared to placebo combined with chemotherapy in first-line treatment of metastatic pancreatic ductal adenocarcinoma (mPDAC) using the Time to Tumor Recurrence evaluated by researchers.
Adverse events | Sign the informed consent form, and until 28 days after the last medication administration
  Evaluate the safety of TQB2868 injection and anlotinib hydrochloride capsules combined with chemotherapy compared to placebo combined with chemotherapy in first-line treatment of metastatic pancreatic ductal adenocarcinoma (mPDAC) by assessing the incidence and severity of adverse events, determined according to the NCI Common Terminology Criteria for Adverse Events (CTCAE) 5.0 grading scale.

CONTACTS AND LOCATIONS:
Locations (70):
- China (70):
  - The First Affiliated Hospital of USTC Anhui Provincial Hospital, Hefei, Anhui
  - Anhui Provincial Cancer Hospital, Hefei, Anhui
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Beijing Friendship Hospital,Capital Medical University, Beijing, Beijing Municipality
  - The Fifth Medical Center of Chinese People's Liberation Army General Hospital, Beijing, Beijing Municipality
  - Beijing Daxing District People'S Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Mengchao Hepatobiliary Hospital OF Fujian Medical University, Fuzhou, Fujian
  - The Firstaffiliated Hospital of Xiamen University, Xiamen, Fujian
  - Zhongshan Hospital Xiamen University, Xiamen, Fujian
  - Gansu Provincial Hospital, Lanzhou, Gansu
  - The First Hospital of Lanzhou University, Lanzhou, Gansu
  - Lanzhou University Second Hospital, Lanzhou, Gansu
  - Sun Yat-Sen University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong
  - Longhua District Central Hospital, Shenzhen, Guangdong
  - Guangxi Cancer Institute, Nanning, Guangxi
  - Guizhou Medical University Affiliated Cancer Hospital Co., LTD, Guiyang, Guizhou
  - Affiliated Hospital of Zunyi Medical Universityl, Zunyi, Guizhou
  - Hainan general hospital, Haikou, Hainan
  - Cancer Hospital Chinese Academy pf Medical Sciences, Langfang, Hebei
  - Tangshan peopel's Hospital, Tangshan, Hebei
  - Daqing Oilfield General Hospital, Daqing, Heilongjiang
  - Harbin Medical University Cancer Hospital, Haerbin, Heilongjiang
  - The First Affiliated Hospital of Henan University of Science & Technology, Luoyang, Henan
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Zhongnan Hospital of Wuhan University, Wuhan, Hubei
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Xiangyang Central Hospital, Xiangyang, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - People's Hospital of Hunan Province, Changsha, Hunan
  - Xiangya Hospital of Central South University, Changsha, Hunan
  - Peking University Cancer Hospital Inner Mongolia Hospital, Hohhot, Inner Mongolia
  - Jiangyin People'S Hospital, Jiangyin, Jiangsu
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Nantong Tumor Hospital, Nantong, Jiangsu
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Jilin Cancer Hospital, Changchun, Jilin
  - The first hospital of Jilin University, Changchun, Jilin
  - Liaoning Cancer Hospital, Shenyang, Liaoning
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - The Second Affiliated Hospital of PLA Air Force Military Medical University, Xi'an, Shaanxi
  - The First Affiliated Hospital of Xi 'An Jiaotong University, Xi'an, Shaanxi
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Linyi people's hospital, Linyi, Shandong
  - Linyi Cancer Hospital, Liyi, Shandong
  - The Affiliated Hospital Of Medical College Qingdao University, Qingdao, Shandong
  - Zhongshan Hospital, Shanghai, Shanghai Municipality
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Shanghai Sixth People's Hospital, Shanghai, Shanghai Municipality
  - Shanghai General Hospital, Shanghai, Shanghai Municipality
  - Shanxi Cancer Hospital, Taiyuan, Shanxi
  - First Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Sichuan Cancer Hospital, Chengdu, Sichuan
  - The Affiliated Hospital of Southwest Medical University, Luzhou, Sichuan
  - Affiliated Hospital of North Sichuan Medical College, Nanchong, Sichuan
  - Tianjin Cancer Hospital Airport Hospital, Tianjin, Tianjin Municipality
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality
  - People's Hospital of Xinjiang Uygur Autonomous Region, Ürümqi, Xinjiang
  - Yunnan Cancer Hospital, Kunming, Yunnan
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital , affiliated with the Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Ningbo Medical Center Lihuili Hospital, Ningbo, Zhejiang
  - Shaoxing People's Hospital, Shaoxing, Zhejiang
  - Wenzhou Medical University Affiliated First Hospital, Wenzhou, Zhejiang